CLINICAL TRIAL: NCT04651556
Title: Comparison Of Intraperitoneal Instillation Of Magnesium Sulphate and Bupivacaine Versus Intravenous Analgesia In Laparoscopic Surgeries In Pediatrics
Brief Title: Intraperitoneal Magnesium Sulphate and Bupivacaine Versus Intravenous Analgesia in Laparoscopic Surgeries in Pediatrics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ibrahim Walash, assistant lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Intraperitoneal anesthesia
Record Dates: First submitted 2020-11-12; First posted 2020-12-03 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Intraperitoneal Magnesium Sulphate in Laparoscope in Pediatrics
Keywords: intraperitoneal, laparoscopic surgeries, pediatrics
MeSH Terms: interventions — Magnesium Sulfate; Bupivacaine; Acetaminophen; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenteral Analgesia (Active Comparator): receive ordinary analgesics via intravenous route as paracetamol (7.5- 10 mg/kg) and ketorolac (0.5 mg/kg).
  Interventions: Drug: paracetamol & ketorolac
- Intraperitoneal instillation (Active Comparator): receive (Magnesium sulphate 40 mg/kg and bupivacaine 4mg/kg) in 30 ml of isotonic 0.9%N.S intra peritoneal at the end of surgery.
  Interventions: Drug: Magnesium Sulfate & bupivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate & bupivacaine — intraperitoneal instillation of a combination of Magnesium sulphate with bupivacaine
  Arms: Intraperitoneal instillation
Drug: paracetamol & ketorolac — parenteral analgesics
  Arms: Parenteral Analgesia

SUMMARY:
The investigators are going to study the analgesic efficacy of intraperitoneal instillation of a combination of Magnesium sulphate with bupivacaine versus ordinary used parenteral analgesics for pain relief after laparoscopic surgeries in pediatrics.

DETAILED DESCRIPTION:
Laparoscopic surgery is a modern surgical technique used for various surgeries such as cholecystectomy, appendectomy and hernia repair. There are a number of advantages of this technique including reduced pain and bleeding, shorter recovery time and hospital stay, and over all reduced healthcare costs. The type of pain after laparoscopic surgery differs considerably from that occurs after laparotomy. Usually patients experience diffuse pain in abdomen, back and shoulder. Acute pain after laparoscopic cholecystectomy has three different components: incisional pain (somatic pain), visceral pain (deep intra-abdominal pain), and shoulder pain (presumably referred visceral pain) . Postoperative nausea and vomiting is a commonly observed phenomenon after laparoscopic procedures. Its incidence increases depending on the anesthetic techniques used. Pain intensity usually peaks during the first postoperative period and usually declines over the following 2-3 days. Pain can prolong hospital stay and lead to increased morbidity.

Inadequately treated pain may lead to splinting, loss of sighing and decrease in vital capacity, and these may contribute to postoperative pulmonary morbidity. Various multimodal approaches have, therefore, been tried to ameliorate postoperative pain. These include parenteral analgesics, local infiltration with local anesthetics, epidural and intrathecal opioids and local anesthetics, interpleural and intercostals nerve blocks as well as intraperitoneal routes that in turn has been explored with local anesthetics and opioids . In order to get an instant relief, polypharmacy is commonly practiced which can be potentially harmful to the patient and can lead to re-admission. It has been appreciated that multiple glutamate receptors are expressed on peripheral nerve terminals, and these may contribute to peripheral nociceptive sensation .

Administration of magnesium sulphate via different routes has been used in anaesthetic practice for decreasing perioperative pain. Parenteral magnesium sulphate has been used for many years as an antiarrhythmic agent and for seizure prophylaxis in eclampsia and preeclampsia. It is N-methyl d-aspartate (NMDA) receptor antagonist and suppresses these receptor induced inflammation and hyper responsiveness . The antinociceptive effect of magnesium sulphate is not only useful in chronic pain, but it also determines in part, the duration and intensity of postoperative pain . These effects are due to calcium antagonism and decrease influx of calcium into the cell and antagonism of NMDA receptor. As these receptors regulate neuronal signalling and are involved in pain processing, magnesium sulphate by blocking this receptor, decreases postoperative pain as well .

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II.
2. Both genders are eligible for study.
3. Patients age from 1 year to 12 years.
4. Patients undergoing laparoscopic surgeries.

Exclusion Criteria:

* 1- ASA III, IV and V class patients. 2- Presence of psychiatric disease. 3- Those with an allergy to any of the study drugs will be excluded from the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
FLACC score | 0 minutes (immediately) postoperative
  (Face, Leg, Activity, Cry, and Consolability) pain assessment score The scale is scored in a range of 0-10 with 0 representing no pain. assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.
FLACC score | 1 hour postoperative
  (Face, Leg, Activity, Cry, and Consolability) pain assessment score The scale is scored in a range of 0-10 with 0 representing no pain. assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.
FLACC score | 6 hours postoperative
  (Face, Leg, Activity, Cry, and Consolability) pain assessment score The scale is scored in a range of 0-10 with 0 representing no pain. assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.
FLACC score | 12 hours postoperative
  (Face, Leg, Activity, Cry, and Consolability) pain assessment score The scale is scored in a range of 0-10 with 0 representing no pain. assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.
FLACC score | 24 hours postoperative
  (Face, Leg, Activity, Cry, and Consolability) pain assessment score The scale is scored in a range of 0-10 with 0 representing no pain. assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.

SECONDARY OUTCOMES:
Vital signs | preoperative, postoperative (0,1,3,6,12,24 hours)
  Heart rate
Vital signs | preoperative, postoperative (0,1,3,6,12,24 hours)
  Arterial blood pressure
Vital signs | preoperative, postoperative (0,1,3,6,12,24 hours)
  Arterial Oxygen saturation
Time to first analgesic administration | 24 hours postoperative
  Time to first analgesic administration
Total analgesic requirements | 24 hours postoperative
  Total analgesic requirements in 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university, Menoufia, Menoufia, Egypt